CLINICAL TRIAL: NCT00496600
Title: Phase I Study of Patupilone and RAD001 in Patients With Refractory Solid Tumor Malignancy
Brief Title: Phase I Study of Patupilone and RAD001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: Novartis Pharmaceuticals (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 050612; CRAD001US16; 0220060307 (Other: CINJ IRB)
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Refractory Malignancy
MeSH Terms: conditions — Neoplasms | interventions — epothilone B; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Patupilone — RAD001 will be taken orally starting at a dose of 30 mg every week for the first cohort of patients, one hour prior to administration of patupilone. Patupilone will then be administered as an infusion, starting at 5 mg/m2 for the first cohort of patients. The dosage and scheduling of RAD001 and patupilone during each 21-day cycle will vary according to cohort assignment
Drug: RAD001 — RAD001 will be taken orally starting at a dose of 30 mg every week for the first cohort of patients, one hour prior to administration of patupilone. Patupilone will then be administered as an infusion, starting at 5 mg/m2 for the first cohort of patients. The dosage and scheduling of RAD001 and patupilone during each 21-day cycle will vary according to cohort assignment

SUMMARY:
This is an unblinded, dose escalation study of patupilone in combination with RAD001 in subjects with advanced cancer to find the maximum tolerated dose of each drug. The purpose of this study is to see what doses of RAD001 and patupilone are safe to use when the two drugs are used at the same time. Other goals in this study are to learn about the effect of RAD 001 and patupilone on tumor growth; to find out what amount of RAD001 is present in the blood when it is combined with patupilone; to learn about proteins in the blood that may predict or show an effect of RAD001 or patupilone and to learn if any changes are seen in the tumor with the type of test called a PET scan.Subjects will be assigned to a dosing group. The dose of patupilone and RAD001 a subject gets depends on when they enter onto this study. The initial subjects in the study will take the lowest doses of RAD001 and patupilone. At least 3 subjects will be treated in each dosing group starting with the smallest dose. If there are few or easy to handle side effects, the next group of at least 3 people to enter in the study will get the next higher dose. This continues until the highest dose of the study drug is found that does not cause serious or hard to treat side effects. Both the subjects and the study doctor will know which dose is assigned. In this study, RAD001 will be given as tablets to take with water. RAD001 will be taken for either 7, 14, or 21 days of each 21 day cycle depending on which dosing group is assigned. If taking RAD 001 and patupilone on the same day, then RAD 001 will be taken with water however prior to receiving patupilone.Patupilone will be given by an intravenous injection (through a vein) for 20 minutes on Days 1 or day 6 of the 21-day cycle. The patupilone dose will be based on height and weight. Blood tests (approximately 1-3 teaspoons) will be done every week. Every six weeks a CT scan or MRI will be done to assess the tumor size. Subjects will continue to receive RAD001 and patupilone as long as the tumor is stable or shrinking, and not having too many side effects from treatment.

DETAILED DESCRIPTION:
Primary Endpoint To identify the maximum tolerated doses (MTD) of the combination of patupilone and RAD001

Secondary Endpoints To assess the toxicity of patupilone and RAD001 To determine if concentrations of RAD001 are elevated in the presence of patupilone To evaluate tumor response using standard imaging modalities (CT scan, x-ray, bone scan) To develop pharmacodynamic markers that may predict or indicate response to mTOR inhibition or patupilone treatment.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have malignancy refractory to standard therapy or for whom no standard, effective therapy is available.
* Patient must have performance status 0-2 on the ECOG Performance Status (see Appendix B)
* Patient's disease must be measurable (RECIST) or evaluable (e.g., cytologically or radiologically detectable disease such as ascites, peritoneal deposits, or lesions which do not fulfill RECIST criteria for measurable disease).
* Patients must have intact intestinal absorption
* Patients must have adequate organ function
* Patient must have recovered from toxicity of prior chemotherapy and/or radiotherapy. Patient may not have received chemotherapy in the prior 4 weeks. Patients may have not received radiotherapy in the prior 3 weeks.
* Patient (male or female) must be ≥ 18 years old.
* Women must not be pregnant or lactating. Female patients of childbearing potential must have a negative pregnancy test within 7 days before initiation of study drug dosing. Post menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male and female patients of reproductive potential must agree to employ an effective barrier method of birth control throughout the study, and for three months following discontinuation of study drug.
* Signed written informed consent.

Exclusion Criteria:

* Patient has received greater than 3 prior cytotoxic regimens for metastatic disease.
* Prior therapy with epothilones, rapamycin, rapamycin analogs, or known sensitivity to these agents
* Prior treatment with any investigational drug within the preceding 4 weeks.
* Patient has history of bone marrow or stem cell transplant.
* Patient has received prior radiation therapy to greater than 25% of the bone marrow.
* Patients has newly diagnosed, not yet treated or uncontrolled brain metastases or leptomeningeal disease.
* Patient has known hypersensitivity to the components of study drugs or its analogs.
* Patient with known Grade 3 or 4 hypersensitivity to macrolide antibiotics (eg. clarithromycin, erythromycin, azithromycin).
* Patient with any active (acute or chronic) or uncontrolled infection requiring systemic therapy.
* Patients with chronic treatment with systemic steroids or another immunosuppressive agent
* Patient with known HIV infection.
* Patients with unresolved diarrhea within the last 7 days prior to start of treatment.
* Concomitant treatment with medications that are listed as clinically relevant inducers or inhibitors of cytochrome P450 (CYP3A).
* Patients taking Coumadin® or other agents containing warfarin, with the exception of low dose Coumadin® (1 mg or less) administered prophylactically for maintenance of in-dwelling lines or ports
* Herbal preparations or related over-the-counter preparations containing herbal ingredients (eg. St. John's Wort)
* Any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as: unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤ 6 months prior to first study treatment, serious uncontrolled cardiac arrhythmia, or severely impaired lung function
* Any patient with uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN
* Any patient with nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with the study therapy
* Patients with liver disease such as cirrhosis, chronic active hepatitis, or chronic persistent hepatitis
* Patients receiving immunization with attenuated live vaccines during study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To identify the maximum tolerated doses (MTD) of the combination of patupilone and RAD001 | 3 years

SECONDARY OUTCOMES:
find toxicity of patupilone and RAD001, see if concentrations of RAD001 are elevated with patupilone, evaluate tumor response using standard imaging, develop pharmacodynamic markers that may predict/indicate response to mTOR inhibition or patupilone trt | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Stein, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- The Cancer Institute of New Jersey, New Brunswick, New Jersey, United States